CLINICAL TRIAL: NCT01693653
Title: Tocilizumab for the Treatment of Behcet's Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment
Sponsor: NYU Langone Health (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-01182
Record Dates: First submitted 2012-09-19; First posted 2012-09-26 (Estimated); Results first posted 2016-06-02 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Behcet Syndrome
Keywords: Behcet's syndrome; oral ulcers
MeSH Terms: conditions — Behcet Syndrome; Oral Ulcer | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tocilizumab (Active Comparator): tocilizumab infusion every 4 weeks over 3 months
  Interventions: Drug: Tocilizumab
- Placebo (Placebo Comparator): placebo infusion 0.9% sodium chloride every 4 weeks over 3 months
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Intravenous infusions every 4 weeks for 3 doses.
  Other Names: actemra

SUMMARY:
This is a double-blind placebo controlled study targeting individuals with active Behcet's Syndrome who have oral ulcers and are resistant (have not responded after 4 weeks) to conventional treatments. Maximum allowable dose of colchicine (0.6mg twice a day) and stable dose for 4 weeks before enrollment. Prednisone or equivalent (< 10mg/day) permitted if dose stable for 6 weeks prior to enrollment.

The study will investigate the safety of tocilizumab for this vasculitic condition in addition to its efficacy.

The planned sample size is 30 participants per arm for a total of 60 participants. The study would be for 3 months, with a safety follow up at 2 months after study termination.

Study participants will stay on their current treatments and either tocilizumab or placebo infusions will be given every 4 weeks in addition. Patients will be randomized to Actemra IV 8mg/kg Q 4 weeks X 3 doses or placebo.

DETAILED DESCRIPTION:
Behcet's syndrome is a vasculitis that causes oral and genital ulcerations, skin lesions, eye disease and arthritis, in addition to vascular complications with thrombophlebitis, thrombosis and rarely central nervous system involvement. IL-6 activity has been suggested in the pathogenesis in some studies. Tocilizumab with its unique mode of action among biologic agents may be a good candidate in this orphan disease.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with BS with at least 1 active oral ulcer resistant (have not responded after 4 weeks to colchicine or local measures.
2. dose (maximum allowable 0.6mg twice a day ) stable for 4 weeks and prednisone or equivalent (maximum dose < 10mg/day) stable for 6 weeks prior to enrollment.
3. Patients must have Behcet's syndrome based on International Study Group criteria.

Patients will be included in the trial based on the following criteria:

* Normal organ function, except if abnormal due to the disease under investigation such as mucocutaneous involvement or joint involvement.
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months after completion of treatment.
* Subject has provided written informed consent.

Exclusion Criteria:

1. Patients with eye, CNS, vascular involvement such as DVT, thrombosis, or aneurysms.
2. Patients who are currently being treated or have been exposed in the last 3 months to other immunosuppressive medications (azathioprine, TNF inhibitors, methotrexate, mycophenolate mofetil). Patients who are currently being treated or have been exposed to Cyclosporine or cyclophosphamide in the past 6 months will be excluded).
3. Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization.
4. Treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational drug, whichever is longer) of screening.
5. Previous treatment with any cell-depleting therapies, including investigational agents or approved therapies, some examples are CAMPATH, anti-CD4, anti-CD5, anti¬CD3, anti-CD19 and anti-CD20 (please note exceptions above).
6. Treatment with intravenous gamma globulin, plasmapheresis or Prosorba column within 6 months of baseline.
7. Immunization with a live/attenuated vaccine within 4 weeks prior to baseline.
8. Previous treatment with TCZ (an exception to this criterion may be granted for single dose exposure upon application to the sponsor on a case-by-case basis).
9. Any previous treatment with alkylating agents such as chlorambucil, or with total lymphoid irradiation.
10. History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies.
11. Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine (include uncontrolled diabetes mellitus) or gastrointestinal disease (including complicated diverticulitis, ulcerative colitis, or Crohn's disease.)
12. Current liver disease as determined by principal investigator unless related to primary disease under investigation
13. Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (including but not limited to tuberculosis and atypical mycobacterial disease, Hepatitis B and C, and herpes zoster, but excluding fungal infections of nail beds).
14. Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening.
15. Active TB requiring treatment within the previous 3 years. Patients should be screened for latent TB and, if positive, treated following local practice guidelines prior to initiating TCZ. Patients treated for tuberculosis with no recurrence in 3 years are permitted. (Appendix 8)
16. Primary or secondary immunodeficiency (history of or currently active) unless related to primary disease under investigation.
17. Evidence of active malignant disease, malignancies diagnosed within the previous 10 years (including hematological malignancies and solid tumors, except basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that has been excised and cured), or breast cancer diagnosed within the previous 20 years unless related to primary disease under investigation.
18. Pregnant women or nursing (breast feeding) mothers.
19. Patients with reproductive potential not willing to use an effective method of contraception.
20. History of alcohol, drug or chemical abuse within 1 year prior to screening.
21. Neuropathies or other conditions that might interfere with pain evaluation unless related to primary disease under investigation.
22. Patients with lack of peripheral venous access.

    Laboratory Exclusion criteria (at screening):
23. Serum creatinine > 1.6 mg/dL (141 µmol/L) in female patients and > 1.9 mg/dL (168 µmol/L) in male patients. Patients with serum creatinine values exceeding limits may be eligible for the study if their estimated glomerular filtration rates (GFR) are >30.
24. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 times upper limit of normal (ULN)
25. Total Bilirubin > ULN
26. Platelet count < 100 x 109/L (100,000/mm3)
27. Hemoglobin < 85 g/L (8.5 g/dL; 5.3 mmol/L)
28. White Blood Cells < 3.0 x 109/L (3000/mm3)
29. Absolute Neutrophil Count < 2.0 x 109/L (2000/mm3)
30. Absolute Lymphocyte Count < 0.5 x 109/L (500/mm3)
31. Positive Hepatitis BsAg, or Hepatitis C antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Yazici, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Center for Musculoskeletal Care, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tocilizumab | Placebo
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tocilizumab | Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Sex/Gender, Customized [Number; unit: participants] | 1 |  | 1
Race/Ethnicity, Customized [Number; unit: particpants] | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome
Description: The study was terminated. No data were collected for this Outcome Measure.
Time Frame: 9 months
Population: The study was terminated. No data were collected for this Outcome Measure.
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Genital Ulcers
Description: The study was terminated. No data were collected for this outcome measure.
Time Frame: 9 months
Population: Terminated due to low enrollments. Data for 1 subject not analyzed.
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Oral Ulcers
Description: The study was terminated. No data were collected for this outcome measure.
Time Frame: 9 months
Population: Terminated due to low enrollments. Data for 1 subject not analyzed.
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Treatment Failures
Description: The study was terminated. No data were collected for this outcome measure.
Time Frame: 9 months
Population: Terminated due to low enrollments. Data for 1 subject not analyzed.
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Oral Ulcer Pain
Description: The study was terminated. No data were collected for this outcome measure.
Time Frame: 9 months
Population: Terminated due to low enrollments. Data for 1 subject not analyzed.
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Gential Ulcer Pain
Description: The study was terminated. No data were collected for this outcome measure.
Time Frame: 9 months
Population: Terminated due to low enrollments. Data for 1 subject not analyzed.
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: BSAS
Description: The study was terminated. No data were collected for this outcome measure.
Time Frame: 9 months
Population: Terminated due to low enrollments. Data for 1 subject not analyzed.
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: MDHAQ
Description: The study was terminated. No data were collected for this outcome measure.
Time Frame: 9 months
Population: Terminated due to low enrollments. Data for 1 subject not analyzed.
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: BDCAF
Description: The study was terminated. No data were collected for this outcome measure.
Time Frame: 9 months
Population: Terminated due to low enrollments. Data for 1 subject not analyzed.
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Safety
Description: The study was terminated. No data were collected for this outcome measure.
Time Frame: 9 moths
Population: Terminated due to low enrollments. Data for 1 subject not analyzed.
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: serious and non serious adverse events were not observed.
Arm/Group | Tocilizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No